CLINICAL TRIAL: NCT00336622
Title: The Efficacy of a Wrist and Hand Splint in Conjunction With Tendon and Nerve Gliding Exercise for the Treatment of Carpal Tunnel Syndrome: A Randomized Clinical Trial
Brief Title: Efficacy of Wrist/Hand Splints and Tendon/Nerve Gliding Exercises for Carpal Tunnel Syndrome: A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Joan C. Rogers, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0402010
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Splints
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Custom-made splint and tendon-nerve gliding exercises Custom-made splint and no tendon-nerve gliding exercises
  Interventions: Device: Splint fabricated by an OT versus an off-the-shelf splint
- Control (Active Comparator): Off-the-shelf splint
  Interventions: Device: Splint fabricated by an OT versus an off-the-shelf splint

INTERVENTIONS:
Device: Splint fabricated by an OT versus an off-the-shelf splint — Experimental:
  Custom-made splint and tendon-nerve gliding exercises Custom-made splint and no tendon-nerve gliding exercises
  Control:
  Control: Off-the-shelf splint and tendon-nerve gliding exercises Off-the-shelf splint and no tendon-nerve gliding exercises
  Other Names: Experimental; Control

SUMMARY:
The purpose of this randomized clinical trial was to examine the efficacy of a splinting (fabricated versus off-the-shelf splint)and exercise (nerve and tendon gliding versus no exercise) interventions to alter the clinical course of Carpal Tunnel Syndrome (CTS). We hypothesized that the fabricated splint with nerve and tendon gliding exercises condition would yield the best functional outcomes at 4 and 8 weeks posttesting.

DETAILED DESCRIPTION:
The purpose of this randomized clinical trial is to examine the efficacy of a splinting and exercise intervention to alter the clinical course of Carpal Tunnel Syndrome (CTS). Specifically, the aims of the study are to test the efficacy of: (1) a splint, positioning the wrist and metacarpal phalange (MCP) joints at 0 degrees in conjunction with tendon and nerve gliding exercises, (2) a splint positioning the wrist and MCP joints at 0 degrees with no exercise (3) a prefabricated wrist cock up splint positioning the wrist at 20 degrees of extension with tendon and nerve gliding exercises, and (4) usual care, a prefabricated wrist cock-up splint positioning the wrist at 20 degrees of extension with no exercise for decreasing symptoms and increasing function in people with clinically diagnosed CTS. The specific hypotheses of the study are:

(1) Subjects randomized to Experimental Condition 1 will perform better than Subjects randomized to Experimental Condition 2; who will perform better than those randomized to Experimental Condition 3, who in turn will perform better than those Subjects randomized to Usual Care. In that order, Subjects will demonstrate a:

1. Significant decrease in CTS symptoms as measured by the Carpal Tunnel Syndrome Symptom Severity Scale at the 4 week Posttest compared to baseline and further decrease at the 8 week Post-Posttest.
2. Significant decrease in upper extremity disability as measured by the Disability of Arm, Shoulder, and Hand (DASH) questionnaire at the 4 week Posttest compared to baseline and further decrease at the 8 week Post-Posttest.
3. Significant increase in functional ability as measured by functional sensibility (Moberg Pick-Up Test), grip strength (dynamometer) and pinch strength (pinch meter) at the 4 week Posttest compared to baseline.

ELIGIBILITY:
Inclusion Criteria: (1) be at least 18 years of age; (2) have positive Tinels, Phalens, and complaints of nocturnal numbness and tingling. (3) English speaking. The exclusion criteria are; (1) have been diagnosed with a neuropathy other than CTS in the past year (2) pregnant (3) have had a steroid injection into the carpal canal in the past 3 months (4) have thenar atrophy (5) have had a prior carpal tunnel release.

Exclusion Criteria: Pregnant women will be excluded from the study. There is an increased incidence of CTS in pregnant women; however symptoms usually decrease after pregnancy. Thus, it would be difficult to determine if the intervention was effective or if the symptoms resolved after the birth of the child. The physician will rule out pregnancy by patient report. Also, no minors will be included in this study because CTS is not a diagnosis common to minors.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Carpal Tunnel Syndrome Symptom Severity & Functional Status Scale | Pre-Post
  Self-report tool

CONTACTS AND LOCATIONS:
Overall Officials: Teresa L. Brininger, PhD, Principal Investigator — U.S. Army, University of Pittsburgh